CLINICAL TRIAL: NCT04128644
Title: Thoughts and Health - Preventing Depression in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-03347
Record Dates: First submitted 2019-10-03; First posted 2019-10-16 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Depression; Adolescent Development; Mental Disorder, Child
Keywords: depression; prevention; school
MeSH Terms: conditions — Depression; Neurodevelopmental Disorders | interventions — Health; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care+Thoughts & health (Other): 12 sessions of Thoughts & Health. Baseline questionnaires and follow up assessments
  Interventions: Behavioral: Thoughts & health; Other: Treatment as Usual
- Standard of care (Other): Baseline questionnaires and follow up assessments, intervention as usual Student Health
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Thoughts & health — 12 sessions of Thoughts & Health. Baseline questionaires and follow up assessments
  Arms: Standard of care+Thoughts & health
Other: Treatment as Usual — Baseline questionnaires and follow up assessments, intervention as usual, Student Health

SUMMARY:
This study aims to test the feasibility of implementing an Icelandic cognitive-behavioral program designed to prevent depression, called "Thoughts and Health" in a Swedish school setting. The investigators will also evaluate whether implementation of the program has an impact on the participating students, regarding both their mental health and their success in finishing junior high school with passing grades.

DETAILED DESCRIPTION:
Clinical depression is a crucial problem among adolescents. In eighth grade more than half of all students experience headaches, stomach pain, stress, feeling down, and difficulties sleeping. Adolescents affected by depression at a young age are at greater risk of experiencing depressive symptoms as adults, with serious impacts on their quality of life and ability to work. Recent reports from the National Board of Health and Welfare have shown that depression is increasing among adolescents and there is now focus on implementing practice-oriented preventative programs for youth.

Studies by members of our research team have shown that a cognitive-behavioral, developmentally-based intervention program, called "Thoughts and Health", prevented initial episodes of depression and/or dysthymia in adolescents for up to 12 months after program completion.

This study aims to test the feasibility of implementing that program in a Swedish school setting, while also collecting and analyzing preliminary results regarding the potential impact of the program on number of students developing depressive symptoms and the number passing junior high school with full grades.

This is an intervention study with a control group. Students from two Swedish junior high schools will be identified as "at-risk" and invited to participate in the program (n=40), while students from two other schools will act as controls (n=40). All participating students will be followed from study start (baseline) and 1, 6, 12, and 18 months after program completion. Results will include quantitative clinical measures, qualitative focus group discussions, and students' final grades. Two courses of the program will be run over two school years. This study involves close collaboration between academia, primary care, and the community.

This is to our knowledge the first study in Sweden that employs a longitudinal design to evaluate the effects of a school program aimed at preventing depression in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Eight grader (school)
* Completed Childrens Depression Inventory (CDI) screening
* Able to understand Swedish both orally and written to a level that he/she can complete forms and questionnaires by themselves

Exclusion Criteria:

* Current or past depression
* Unable to function in a group session
* Current psychotherapeutic treatment
* Past or current suicidal thoughts or attempts

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Depressive episode | 18 months
  Number of participants that have scores that indicate a depressive episode. Questionnaire CDI (Children Depression Inventory), CDI has 27 items scores, each item range from 0-3, above the 90th percentile indicate depressive problems, 90th percentile indicate depressive episode.

SECONDARY OUTCOMES:
Complete grades | 18 months
  Measures if participants have complete grades from ninth grade when finishing school. Will be collected through public school registers.

OTHER OUTCOMES:
Life quality | 18 month
  Collect data from participants through questionnaire: MHC- SF (Mental health continuum), MHC-SF consists of 14 items asking about the frequency of experiences the last month. There are three items on emotional well-being such as feelings of being happy, interested in life and satisfied, five items on social well-being referring to acceptance, actualization, contribution, coherence and integration and six items on psychological well-being capturing purpose in life, environmental mastery, autonomy, personal growth, positive relations and self-acceptance. Answers are given on a 6-point Likert scale from 0-6.
Social adjustment | 18 month
  Collect data from participants through questionnaire: EWSAS (Education Work Social Adjustment Scale), EWSAS consists of 5 items asking if and to what amount the mental health issues are affecting friendships, family relationships, school environment and social activities. Likert scale from 0-8.
Mental health | 18 month
  Collect data from participants through questionnaire: RCADS (Revised Anxiety and Depression Scale), It is designed to assess clinical syndromes of anxiety as well as depression, building on the DSM-IV criteria. The RCADS provides two total scores, and 6 subscales: Separation Anxiety Disorder (SAD), Social Phobia (SoP), Obsessive Compulsive Disorder (OCD), Panic Disorder (PD), (GAD) and Major Depressive Disorder (MDD). The higher the score the more symptoms of mental health issues. The scale grades from 0-141.
Mental Clinical Assessment | 18 month
  Assessment through Clinical interview: MINI-KID (Mini International Neuropsychiatric Interview)

CONTACTS AND LOCATIONS:
Overall Officials: Josefine Lilja, PhD, Principal Investigator — Vastra Gotaland Region
Locations (1):
- FoU Research and Development, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Immediately following publication, individual participant data that underlie the result, after de-identification (text, tables, figures, and appendices) will be available. Researchers that provide a sound and methodological proposal will gain access to achieve aims in the approved proposal. Proposals should be directed to josefine.lilja@vgregion.se To gain access, data requestor s will need to sign a data access agreement.
Supporting Information: Study Protocol, ICF
Time Frame: After publication of long term follow up (18month follow up) and then no end date.

REFERENCES:
- [Derived] Wikberg C, Augustsson P, Sveinsdottir G, Craighead WE, Arnarson EO, Marteinsdottir I, Lilja JL. Is the Thoughts and Health programme feasible in the context of Swedish schools? A quasi-experimental controlled trial study protocol. BMJ Open. 2021 Jan 22;11(1):e040374. doi: 10.1136/bmjopen-2020-040374. PMID 33483440